CLINICAL TRIAL: NCT04038931
Title: Collection of Human Liver Biopsy and Whole Blood Samples From Type 1 Diabetes Mellitus (T1DM), Total or Partial Pancreatectomy Patients for Potential Use as an Autologous Source for Insulin Producing Cells in Future Clinical Studies
Brief Title: Collection of Human Liver Biopsy and Whole Blood Samples From T1DM, TP or PP Patients for Potential Use for Insulin Producing Cells in Future Clinical Studies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Orgenesis Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ORG-ISR-01
Record Dates: First submitted 2019-06-03; First posted 2019-07-31 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes; Pancreatectomy; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Liver biopsy collection — Liver biopsy collection to Confirm suitability of T1DM, total or partial pancreatectomy patient's liver cells to be used as future personalized cell replacement therapy.

SUMMARY:
In this study, liver samples will be collected, processed and stored in a specialized, clinical grade, cell bank for potential future clinical use. A set of ex-vivo immunogenicity and transdiffrentiation tests will be carried to confirm the ability of this cryopreserved cell batch to be used as clinical grade raw material. Biopsies will be collected during TP or PP with the assumption that some of the patients (especially PP patients will not go through Islets autotransplantation) will develop brittle diabetes, thus Orgenesis therapy can provide them in the long run, a treatment. In terms of T1DM the purpose is to have available clinical grade raw material for cell replacement therapy.

The collected liver samples will be proliferated (up to passage 4) for future use. A portion of the stored cells will be utilized in a small-scale process to test possible immunogenicity performed on the collected blood sample. The assay will provide data whether immunomodulation treatment will be required in the future clinical trials. Also the transdffrentiated cells (AIPs) will be tested according to release criteria relevant for clinical IPC production. Liver biopsy donors will be contacted upon approval of the consecutive study and will have study recruitment priority. The donors can refuse to participate in the future study or may not need the therapy, however, their biopsies will be stored for a potential use if required, after the therapy is approved.

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 18 and 70 years old, inclusive.
* For T1DM - Patients with history of established T1DM undergoing an elective abdominal surgery with an easy access to the liver
* Patients undergoing total or partial Pancreatectomy
* Female patients who agree not to breastfeed during the study up to at least seven days after the study is completed.
* For T1DM - Receiving multiple daily insulin injections or insulin pump therapy.
* For T1DM - HbA1c ≤10%.
* Willing to sign the study informed consent document.
* In good general health with no infections, or concomitant medical conditions that would influence the outcome of the trial, at the discretion of the Investigator and the Sponsor.

Exclusion Criteria:

* Received any investigational product within 30 days of admission into this study or plan to participate in any other clinical study during the conduct of this study.
* Received methotrexate or other rheumatoid disease modifying agents within the last 6 months.
* Administration of a live vaccine 30 days prior to screening.
* No evidence of liver Cirrhosis or Nonalcoholic Steatohepatitis (NASH, grade 3 and above) within the last month.
* Patients diagnosed with liver viral infections such as HBV, HCV, HIV
* Patients diagnosed with CMV (defined by IgM positive).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study population comprises of patients undergoing total or partial pancreatectomy or from T1DM patients undergoing an elective abdominal surgery (in which there is an easy access to the liver).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-06-20 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
Confirmation of patients' suitability eligibility to participate in future clinical study | 1 year post biopsy collection
  Defined by a successful AIPs production from their liver biopsy.
Evaluating autoimmune response to AIPs | 1 year post biopsy collection
  Defined by Mixed Lymphocyte Reaction (MLR) assay based on the patient's PBMCs isolated from whole blood samples and following in-vivo subcutaneous implantation into the patients' arm